CLINICAL TRIAL: NCT00537303
Title: Comparison of the Efficacy and Safety of Step-wise Addition of Short Acting Insulin Analogue Insulin Aspart to Once Daily Insulin Detemir and Oral Anti-diabetic Treatment in Patients With Type 2 Diabetes
Brief Title: Comparison of the Blood Sugar Lowering Effect and Safety of Two Insulin Treatments in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1833; 2007-000123-18 (EudraCT Number)
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Results first posted 2010-08-13 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advanced (Experimental): Insulin detemir once daily + oral anti-diabetic drugs (OADs) with addition of meal-time insulin aspart stepwise (1-2-3) at the meals with the largest prandial increments and individually adjusted insulin aspart based mainly on postmeal SMPG (self monitored plasma glucose). The stepwise addition occurred if the treatment target of HbA1c below 7.0% was not reached after 12, 24 and 36 weeks, respectively.
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- Basic (Active Comparator): Insulin detemir once daily + oral anti-diabetic drugs (OADs) with addition of meal-time insulin aspart stepwise (1-2-3) at the largest meals and individually adjusted insulin aspart based mainly on pre-meal and bedtime SMPG (self monitored plasma glucose). The stepwise addition occurred if the treatment target of HbA1c below 7.0% was not reached after 12, 24 and 36 weeks, respectively.
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target dose titration scheme (individually adjusted dose) for a once daily injection s.c. (under the skin)
Drug: insulin aspart — Administered 1 - 3 times daily, at largest prandial increment, injection s.c. (under the skin)
  Arms: Advanced
Drug: insulin aspart — Administered 1 - 3 times daily, at largest meals, injection s.c. (under the skin)
  Arms: Basic

SUMMARY:
This trial is conducted in Europe, Africa and the United States of America (USA).

The aim of this trial is to compare the safety and efficacy of two different insulin treatments, the "basic" and the "advanced" treatment in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus for more than 6 months
* HbA1c (glycosylated haemoglobin A1c) between 7.5 % and 10.0% at trial initiation (screening)
* BMI (Body Mass Index) less than 40 kg/m2
* Basal insulin treatment for at least 3 months (NPH once or twice daily, insulin glargine or detemir once daily)
* Treatment with one to 3 OADs

Exclusion Criteria:

* Known or suspected allergy to trial products or related products
* Women who are pregnant, are breast-feeding or intend to become pregnant within the next 48 weeks
* Previous participation in any trial including this for the last 6 months
* Use of more than 1 U/kg of basal insulin daily at trial initiation (screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (63):
- United States (18):
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Mission Viejo, California
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Novo Nordisk Investigational Site, Århus C, Denmark
- Finland (5):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Vaasa
  - Novo Nordisk Investigational Site, Vantaa
- France (5):
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Pointe à Pitre
  - Novo Nordisk Investigational Site, Vénissieux
- Netherlands (6):
  - Novo Nordisk Investigational Site, 's-Hertogenbosch
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Etten-Leur
  - Novo Nordisk Investigational Site, Hulst
  - Novo Nordisk Investigational Site, Utrecht
  - Novo Nordisk Investigational Site, Woerden
- Norway (6):
  - Novo Nordisk Investigational Site, Jessheim
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Sarpsborg
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Tromsø
  - Novo Nordisk Investigational Site, Tønsberg
- Novo Nordisk Investigational Site, Moscow, Russia
- Serbia and Montenegro (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Nis
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
- Spain (7):
  - Novo Nordisk Investigational Site, Cáceres
  - Novo Nordisk Investigational Site, Inca
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Mérida
  - Novo Nordisk Investigational Site, Mostoles - Madrid -
  - Novo Nordisk Investigational Site, Santiago de Compostela
- Sweden (3):
  - Novo Nordisk Investigational Site, Ängelholm
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Mölndal
- United Kingdom (7):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, Llanelli
  - Novo Nordisk Investigational Site, Llantrisant
  - Novo Nordisk Investigational Site, Reading
  - Novo Nordisk Investigational Site, Rugby

REFERENCES:
- [Result] Meneghini L, Mersebach H, Kumar S, Svendsen AL, Hermansen K. Comparison of 2 intensification regimens with rapid-acting insulin aspart in type 2 diabetes mellitus inadequately controlled by once-daily insulin detemir and oral antidiabetes drugs: the step-wise randomized study. Endocr Pract. 2011 Sep-Oct;17(5):727-36. doi: 10.4158/EP10367.OR. PMID 21550957
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 centres in 12 countries participated: Denmark (1), Finland (6), France (5), Netherlands (6), Norway (5), Russian Federation (4), Serbia (2), South Africa (3), Spain (5), Sweden (3), United Kingdom (7), United States of America (20)
Pre-assignment Details: Eligible subjects were included in a 12-weeks forced titration period with insulin detemir as add-on to current oral anti-diabetic drug (OAD) treatment. Those subjects who did not meet the HbA1c target below 7% were then randomised to one of the two treatment regimens. Any use of sulphonylurea was discontinued at the time of randomisation.
Period: Overall Study
Arm/Group | Advanced | Basic
Started | 146 | 150
Completed | 120 | 125
Not Completed | 26 | 25
Not completed — Adverse Event | 1 | 4
Not completed — Lack of Efficacy | 6 | 7
Not completed — Protocol Violation | 8 | 4
Not completed — Withdrawal criteria | 3 | 3
Not completed — Unclassified | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advanced | Basic | Total
Number analyzed (Participants) | 146 | 150 | 296
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 117 | 122 | 239
  >=65 years | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.29) | 58.3 (8.54) | 58.3 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 67 | 137
  Male | 76 | 83 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 34 | 60
  Not Hispanic or Latino | 108 | 103 | 211
  Unknown or Not Reported | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 120 | 122 | 242
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 25
Height [Mean (Standard Deviation); unit: meter] | 1.68 (0.10) | 1.67 (0.10) | 1.68 (0.10)
Body weight [Mean (Standard Deviation); unit: kg] | 88.8 (15.8) | 88.0 (16.3) | 88.4 (16.0)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 31.26 (4.26) | 31.38 (4.92) | 31.32 (4.60)
Stratification [Number; unit: participants]
  Metformin alone | 62 | 64 | 126
  Metformin + other OAD | 84 | 86 | 170
HbA1c (glycosylated haemoglobin A1c) [Mean (Standard Deviation); unit: percentage (%) of total haemoglobin] | 8.89 (1.16) | 8.67 (0.97) | 8.78 (1.07)
Diabetes history [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 11.82 (5.99) | 12.68 (6.68) | 12.25 (6.35)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: Analysed for the full analysis set.
Time Frame: week 36
Population: Full analysis set (FAS) is all randomised subjects exposed to at least one dose of trial products.
Measure: Least Squares Mean (Standard Error); unit: percentage (%) of total haemoglobin
Arm/Group | Advanced | Basic
Number analyzed (Participants) | 140 | 147
percentage (%) of total haemoglobin | 7.67 (0.09) | 7.61 (0.08)
Statistical Analysis 1: Comparison: Advanced vs Basic; Equivalence analysis with a null hypothesis stating that there is a difference between Advanced and Basic treatment groups of more than 0.4%; Test type: Non-Inferiority or Equivalence — The two treatments are declared equivalent if the 95% Confidence Interval for the estimated difference in means between the two treatment groups is included in the interval from -0.4 to 0.4 for both the full analysis set and the per protocol set; p = 0.606, ANCOVA — P-value for test of difference between treatments; Regimen, country and previous oral antidiabetic drug (OAD) use as factors and baseline HbA1c as covariate; Mean Difference (Final Values) = 0.06, 95% CI [-0.17 to 0.29]

2. Primary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: Measured for the Per Protocol analysis set.
Time Frame: week 36
Population: Per Protocol analysis set: All exposed subjects who completed the trial without significantly violating the inclusion/exclusion criteria or other aspects of the protocol considered to potentially affect the efficacy results.
Measure: Least Squares Mean (Standard Error); unit: percentage (%) of total haemoglobin
Arm/Group | Advanced | Basic
Number analyzed (Participants) | 107 | 118
percentage (%) of total haemoglobin | 7.55 (0.09) | 7.52 (0.08)
Statistical Analysis 1: Comparison: Advanced vs Basic; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.816, ANCOVA — P-value for test of difference between treatments; Mean Difference (Final Values) = 0.03, 95% CI [-0.21 to 0.26]

3. Secondary Outcome: Hypoglycaemic Episodes
Description: Number of hypoglycaemic episodes from Week 0 to Week 36, defined as major, minor or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L (56 mg/dL). Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Weeks 0-36
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial products.
Measure: Number; unit: episodes
Arm/Group | Advanced | Basic
Number analyzed (Participants) | 146 | 150
episodes
  Major | 1 | 4
  Minor | 531 | 567
  Symptoms Only | 283 | 344

4. Secondary Outcome: Biochemistry: Serum Alanine Aminotransferase
Description: Alanine aminotransferase was measured in serum at week 36. Serum samples were analysed at a central laboratory.
Time Frame: week 36
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial products.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Advanced | Basic
Number analyzed (Participants) | 133 | 138
U/L | 30.09 (18.54) | 27.04 (14.64)

5. Secondary Outcome: Haematology: Haemoglobin Measured in Blood
Description: Haemoglobin was measured in blood samples at week 36. Blood samples were analysed at a central laboratory.
Time Frame: week 36
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial products.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Advanced | Basic
Number analyzed (Participants) | 128 | 136
mmol/L | 8.57 (0.87) | 8.58 (0.95)

6. Secondary Outcome: Cardiovascular Risk Marker: High-sensitivity C-reactive Peptide
Description: High-sensitivity C-reactive peptide was measured in serum at week 36. Serum samples were analysed at a central laboratory.
Time Frame: week 36
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial products.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Advanced | Basic
Number analyzed (Participants) | 132 | 136
mg/L | 3.76 (3.46) | 4.67 (6.86)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timeframe of 36 weeks.
Description: Safety analysis set is all randomised subjects exposed to at least one dose of trial products.
Arm/Group | Advanced | Basic
Serious Adverse Events (participants affected / at risk) | 4/146 | 8/150
Other Adverse Events (participants affected / at risk) | 54/146 | 58/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced (N=146) | Basic (N=150)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic Foot Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced (N=146) | Basic (N=150)
Nasopharyngitis (Infections and infestations) | 21 (24) | 17 (22)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 5 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (8)
Headache (Nervous system disorders) | 13 (19) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (8)
Hypertension (Vascular disorders) | 8 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.